CLINICAL TRIAL: NCT07233603
Title: Comparison of the Effects of Subcostal Transversus Abdominis Plane Block Versus Rectus Sheath Block on Postoperative Pain in Midline Abdominal Incision Laparotomy
Brief Title: S-TAP vs RSB in Midline Abdominal Incision Laparotomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Oguz Gundogdu, Associate Professor, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-03/01
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain; Laparotomy
Keywords: postoperative pain; regional anesthesia; laparotomy; midline incision; subcostal transversus abdominis plane block; rectus sheath block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-TAP (Active Comparator): For this group, S-TAP blocks will be performed bilaterally right after the surgery completion with the patients in supine position. For S-TAP, a high frequency linear transducer USG is placed below the xiphoid process, on the linea alba transversely. The probe will then be moved laterally along the costal margin with a slight oblique motion to match the costal arc until the transversus abdominis muscle is visualized under the rectus abdominis muscle. The block needle will be inserted in-plane from inferolateral to superomedial direction, aiming toward the fascial plane between transversus abdominis and rectus abdominis muscles. After negative aspiration and hidrodissection with 1-2 mL of saline and verifying the location of the needle tip, 20 mL of 0.25% bupivacaine will be administered on each side, with a total of 40 mL bilaterally.
  Interventions: Procedure: Subcostal Transversus Abdominis Plane Block
- RSB (Active Comparator): For this group, RS blocks will be performed bilaterally right after the surgery completion with the patients in supine position. For RSB, a high frequency linear transducer USG is placed above the umbilicus transversely. The probe will then be moved laterally until the rectus abdominis muscle, its posterior sheath and the peritoneum can be visualized clearly. The block needle will be inserted in-plane from lateral to medial direction, aiming toward the posterior sheath of the rectus abdominis muscle. After negative aspiration and hidrodissection with 1-2 mL of saline and verifying the location of the needle tip, 20 mL of 0.25% bupivacaine will be administered on each side, with a total of 40 mL bilaterally.
  Interventions: Procedure: Rectus Sheath Block

INTERVENTIONS:
Procedure: Subcostal Transversus Abdominis Plane Block — 20 mL of 0.25% bupivacaine on each side
  Arms: S-TAP
Procedure: Rectus Sheath Block — 20 mL of 0.25% bupivacaine on each side
  Arms: RSB

SUMMARY:
The aim is to compare the postoperative analgesic effects of Subcostal Transversus Abdominis Plane Block (S-TAP) versus Rectus Sheath Block (RSB) in patients undergoing laparotomy with midline abdominal incision.

DETAILED DESCRIPTION:
Patients were divided into two randomized groups: Group 1 (S-TAP group, n=30) and Group 2 (RSB group, n=30). All patients will receive the same standard general anesthesia per hospital protocol. All blocks will be applied with the same ultrasonography and block equipment, and by the same physician. All patients will receive Paracetamol 1gr and Dexketoprofen 50mg intravenous (IV) 10 minutes prior to skin closure. After the surgery was completed, patients in Group 1 will receive subcostal transversus abdominis plane block (S-TAP) with 20 mL of 0.25% bupivacaine bilaterally (with a total volume of 40 mL). Patients in Group 2 will receive rectus sheath block (RSB) with 20 mL of 0.25% bupivacaine bilaterally (with a total volume of 40 mL). Routine analgesic procedure consisting of 3x1gr Paracetamol and 2x50mg Dexketoprofen will be followed postoperatively for 24 hours. Numeric Rating Scale (NRS) will be used to assess postoperative pain on 1st, 6th, 12th, 18th and 24th hours after the surgery. Tramadol 50mg IV will be administered as a rescue analgesic for all patients if NRS score is equal to or higher than 4. Total Tramadol consumption will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients older than 18 years of age who underwent laparotomy with midline incision under general anesthesia and were American Society of Anesthesiologists (ASA) I-II-III according to the ASA risk classification.

Exclusion Criteria:

* patients who did not give consent,
* patients with coagulopathy,
* patients with signs of infection at the block application site,
* patients using anticoagulants,
* patients with local anesthetic drug allergies,
* patients with unstable hemodynamics,
* patients who could not cooperate during postoperative pain assessment
* patients who received ileostomy or colostomy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) Scores | Postoperative 24 hours
  Numerical rating scale is used for pain assessment. The scores of the numerical rating scale changes between 0 to 10 points. 10 points mean "the most severe pain that the patient ever had". 0 point means "there is no pain." Higher scores mean worse outcome.
Total tramadol consumption | Postoperative 24 hours
  Postoperative total rescue analgesic need was recorded as "milligram" in unit.

CONTACTS AND LOCATIONS:
Overall Officials: Oğuz Gündoğdu, Principal Investigator — Sivas Cumhuriyet University School of Medicine, Anesthesiology and Reanimation
Locations (1):
- Sivas Cumhuriyet University, Sivas, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No